CLINICAL TRIAL: NCT01039597
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of the Safety and Therapeutic Activity of ORE1001 in Subjects With Ulcerative Colitis
Brief Title: Safety and Activity of ORE1001 in Subjects With Ulcerative Colitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ore Pharmaceuticals, Inc. (Industry)
Responsible Party: Senior Vice-President of Clinical Development, Ore Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORX102
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Mild to Moderate Ulcerative Colitis
Keywords: IBD; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — 2-(1-carboxy-2-(3-(3,5-dichlorobenzyl)-3H-imidazol-4-yl)ethylamino)-4-methylpentanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active study drug (Experimental): ORE1001 300 mg oral capsules
  Interventions: Drug: ORE1001
- Placebo control (Placebo Comparator): 300 mg oral capsules containing placebo material
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORE1001 — Oral capsules containing 300 mg of the active, study drug
  Other Names: GL1001
  Arms: Active study drug
Drug: Placebo — placebo capsules
  Other Names: matched placebo
  Arms: Placebo control

SUMMARY:
A clinical trial is being conducted to test the effects of a potential new treatment in patients with ulcerative colitis. Study participants will be given capsules containing either ORE1001 or a matching placebo capsule and will take the medicine by mouth for six weeks. Study participants will be asked to visit clinic sites where they will be asked questions about their ulcerative colitis. Small samples of blood will be be drawn at study visits to monitor the participant's health and a tiny sample of tissue will be taken in an endoscopy at two times to determine whether the disease is getting better or worse.

DETAILED DESCRIPTION:
This is a Phase Ib/IIa prospective, multicenter, double blind, randomized, placebo controlled, clinical study to evaluate the safety, tolerability and pilot therapeutic activity of ORE1001, administered as capsules by mouth, for 6 weeks in subjects with Ulcerative Colitis.

Eligible subjects will be randomly assigned to either ORE1001 or placebo, respectively. Sigmoidoscopies with biopsies will be performed at the first treatment visit and week 6.

Subjects will be instructed to self-administer the study drug on an outpatient basis and will be scheduled to return for clinical evaluation on weeks 2, 4, 6 and between Weeks 10-12.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a documented diagnosis of mild to moderate Ulcerative Colitis, as demonstrated clinically and by endoscopy at Visit 2.
2. Baron score greater than or equal to 2 at baseline.
3. Truelove-Witt (modified) score of 14 or less.
4. At least 6 months duration of disease
5. At baseline the subject should have either stable disease or stable disease requiring 5-ASA treatment
6. If on a 5-ASA treatment, subject must have been on stable dose for at least two weeks prior to screening and is expected to continue on that dose until the study is completed
7. Subject has normally functioning major organ systems (aside from gastrointestinal tract) as indicated by medical history, vital signs, physical exam and clinical laboratories (including hematology, coagulation, chemistries and urinalysis).
8. Male or female subjects 18-70 years old
9. Subject has provided voluntary written informed consent to participate in this study.
10. Subject may be of child-bearing potential, but is not pregnant, nursing, or planning a pregnancy for the duration of the study and has a negative pregnancy test prior to enrollment.
11. Subject agrees to use a medically-acceptable form of contraception from screening through 30 days after the final dose of study drug. Female partners of male subjects enrolled into this study are also recommended to use an acceptable method of birth control. Males must agree to not donate sperm during the entire study and for 90 days after the last dose of study drug.

Exclusion Criteria:

1. A clinically significant medical history, medical finding or an ongoing medical or psychiatric condition which, in the opinion of the Investigator, could jeopardize the safety of the subject, impact the validity of the study results, or interfere with the completion of treatment according to this protocol.
2. Subject has an ALT or serum creatinine greater than 1.5 times the upper limit of normal range for the reference lab at screening.
3. Subject who, in the opinion of the investigator, is febrile at screening.
4. Subject had used the following treatments for IBD: steroids or any or biologic immunomodulators or any topical treatments (e.g. enemas) within the last 4 weeks prior to baseline, immunosuppressants or antimetabolites within the preceding 6 weeks, antibiotic use within the previous 7 days or chronic use of any anti-inflammatory drugs (except aminosalicylates) within 7 days.
5. History of illicit drug abuse or positive urine screen for drugs of abuse or history of alcohol abuse if acknowledged at the screening visit or noted in the subject's medical record at screening.
6. Subject has a positive blood screen for HIV, Hepatitis B (HBsAg), or Hepatitis C.
7. Subject has evidence of infectious colitis, e.g., Clostridium difficile, Amoebiasis, Giardia lamblia by stool examination of at screening.
8. Subject has evidence for gastrointestinal parasites as per stool ova and parasites testing at screening.
9. Subject has evidence of tuberculosis by blood interferon gamma release assay at screening.
10. Any uncontrolled, intercurrent illness (e.g., active infection).
11. History of gastrointestinal cancer.
12. Abdominal surgery or any major surgery within the preceding 28 days of the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of ORE1001 in subjects with ulcerative colitis as demonstrated by the frequency and severity of adverse events | 6 Week

SECONDARY OUTCOMES:
Change in the modified Baron Score from Baseline to Week 6 | 6 Week
Change in the Ulcerative Colitis Clinical Score from Baseline | 6 Week
Change in the partial Mayo Score fom baseline | 6 week
Calprotectin concentrations | 6 week
Riley Acute Inflammation Scale (histology) | 6 week
Clinical remission | Week 6

CONTACTS AND LOCATIONS:
Locations (7):
- Robarts Research Institute, London, Ontario, Canada
- India (6):
  - Dr, Bhatnagar's Clinic, Ahmedabad, Gujarat
  - Vikram Jyoth Centre for Advanced Gastroenterology, Mysore, Karnataka
  - St. John's Medical College Hospital, Bangalore, Karnatka
  - Gut-n-HEPA Care, Indore, Madhya Pradesh
  - Amol Gastroenterology Hospital, Indore, Madhya Pradesh
  - B.Y.L. Nair Hospital, Bombay, Maharashtra

REFERENCES:
- [Background] Byrnes JJ, Gross S, Ellard C, Connolly K, Donahue S, Picarella D. Effects of the ACE2 inhibitor GL1001 on acute dextran sodium sulfate-induced colitis in mice. Inflamm Res. 2009 Nov;58(11):819-27. doi: 10.1007/s00011-009-0053-3. Epub 2009 Jun 11. PMID 19517214
- See also: Colitis and Crohn's Foundation of America — http://www.ccfa.org